CLINICAL TRIAL: NCT06573814
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Efficacy of Bio Gelee Royale Forte on Immune Health in Healthy Adults
Brief Title: The Effects of Bio Gelee Royale Forte on Immune Health in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medex d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24MDCFR01
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Upper Respiratory Tract Infection; URTI
Keywords: Upper Respiratory Tract Infection; Safety and efficacy; Royal Jelly
MeSH Terms: conditions — Respiratory Tract Infections | interventions — royal jelly

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bio Gelee Royale Forte (Experimental): Participants will be instructed to take two capsules of study product in the morning on empty stomach once per day for 98 days. If there is an incidence of URTI between enrollment and Day-14, participant will be instructed to start study product intake three days after symptom resolution. If a dose is missed participants are instructed to take the dose approximately two hours after a meal. Participants will be advised not to exceed two capsules daily.
  Interventions: Dietary Supplement: Bio Gelee Royale Forte
- Placebo (Placebo Comparator): Participants will be instructed to take two capsules of study product in the morning on empty stomach once per day for 98 days. If there is an incidence of URTI between enrollment and Day-14, participant will be instructed to start study product intake three days after symptom resolution. If a dose is missed participants are instructed to take the dose approximately two hours after a meal. Participants will be advised not to exceed two capsules daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bio Gelee Royale Forte — Two capsules of Bio Gelee Royale Forte will be taken in the morning on empty stomach once per day for 98 days.
  Other Names: Royal Jelly
  Arms: Bio Gelee Royale Forte
Other: Placebo — Two capsules of placebo will be taken in the morning on empty stomach once per day for 98 days.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Bio Gelee Royale Forte compared to placebo on frequency, severity, and duration of upper respiratory tract infections (URTIs) among adults who are otherwise healthy but susceptible to URTIs during cold and flu season. Additionally, the safety and tolerability of Bio Gelee Royale Forte, as compared to placebo, will be measured by the occurrence of and/or changes in treatment emergent adverse effects.

DETAILED DESCRIPTION:
The investigational product (IP), Bio Gelee Royale Forte, contains royal jelly which is secreted by the hypopharyngeal and mandibular glands of nurse bees. Royal jelly is commonly used as a functional food due to its antibacterial, anti-oxidant, anti-inflammatory, and anti-aging properties. While current evidence suggests royal jelly may play a role in improving human health, little is known about the effects of royal jelly on immune function. Therefore, the objective of this study is to investigate the efficacy of Bio Gelee Royale Forte compared to placebo on immune health in a healthy adult population with self-reported susceptibility to URTIs during cold and flu season.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18-65 years of age, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must self-report confirmation they are not pregnant, do not plan to become pregnant, and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence
3. At least two self-reported incidences of URTI in the last 12 months
4. Agrees to maintain current lifestyle as much as possible throughout the study, including diet, exercise, and sleep
5. Agrees to maintain medications/supplements (particularly those used for immunity support) as much as possible throughout the study and not add new supplements to their routine
6. Able and willing to complete all study assessments
7. Provided voluntary and informed consent to participate in the study
8. Generally healthy as determined by medical history with no unstable diagnosed medical conditions

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of investigational product or placebo ingredients
3. Self-reported allergy to bees or other insects
4. Self-reported autoimmune disease or are immune compromised due to other factors
5. Self-reported current or anticipated severe environmental allergies during the study period requiring medication or need for allergy shots
6. Self-reported ongoing diagnosis of acute or chronic respiratory illness (e.g., asthma, chronic bronchitis, sinusitis, pharyngitis, chronic obstructive pulmonary disease (COPD))
7. Self-reported ongoing and unstable diseases/conditions in the past three months, including:

   1. Arthritis and joint diseases
   2. Gastrointestinal diseases
   3. Hypertension
   4. Type I or type II diabetes
   5. Cardiovascular disease
   6. Kidney diseases
   7. Liver diseases
   8. Thyroid condition
8. Self-reported surgery in the past three months or individuals who have planned surgery during the course of the study
9. Self-reported cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
10. Alcohol intake average of >2 standard drinks per day
11. Alcohol or drug abuse within the last 12 months that has required treatment
12. Current use of prescribed and/or over-the-counter (OTC) medications/supplements that may impact the efficacy and/or safety of the investigational product
13. Participation in other clinical research studies 30 days prior to screening
14. Individuals who are unable to give informed consent
15. Any other condition or lifestyle factor that may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The difference in frequency, severity, and duration of upper respiratory tract infections (URTI). | Day -14 to day 84
  The difference in frequency, severity, and duration of URTIs as assessed by the Wisconsin Upper Respiratory Symptom Survey-24 (WURSS-24) questionnaire over the 84-day supplementation period between Bio Gelee Royale Forte and Placebo. The average severity score of each symptom is scored on scale of 0- no symptom to 7-severe symptom. A higher score would indicate worse outcome.

SECONDARY OUTCOMES:
The difference in frequency of URTIs from day -14 to day -1. | day -14 to day -1
  The difference in frequency of URTIs from day -14 to day -1 as assessed by the WURSS-24 questionnaire, will be compared between Bio Gelee Royale Forte and Placebo.
The difference in frequency of URTIs from day -14 to day 84. | day -14 to day 84
  The difference in frequency of URTIs from day -14 to day -1 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
The difference in severity of URTI symptoms from day -14 to day -1. | day -14 to day -1
  The difference in severity of URTIs from day -14 to day -1 as assessed by the WURSS-24 questionnaire and determined by the average severity scores of URTI symptoms will be compared between Bio Gelee Royale Forte and Placebo.
The difference in severity of URTI symptoms from day -14 to day -1. | day -14 to day -1
  The difference in severity of URTIs from day -14 to day -1 as assessed by the WURSS-24 questionnaire and determined by the area under the curve (AUC) for daily total symptom scores will be compared between Bio Gelee Royale Forte and Placebo. Area under the curve (AUC) for URTI symptoms from WURSS-24 is calculated daily from day -14 to day -1.
The difference in severity of URTI symptoms from day -14 to day 84. | day -14 to day 84
  The difference in severity of URTIs from day -14 to day 84 as assessed by the WURSS-24 questionnaire and determined by the average severity scores of URTI symptoms will be compared between Bio Gelee Royale Forte and Placebo.
The difference in severity of URTI symptoms from day -14 to day 84. | day -14 to day 84
  The difference in severity of URTIs from day -14 to day 84 as assessed by the WURSS-24 questionnaire and determined by the area under the curve (AUC) for daily total symptom scores will be compared between Bio Gelee Royale Forte and Placebo.
The difference in duration of URTI symptoms from day -14 to day -1. | day -14 to day 84
  The difference in duration of URTIs from day -14 to day -1 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
The difference in duration of URTI symptoms from day -14 to day 84. | day -14 to day 84
  The difference in duration of URTIs from day -14 to day 84 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
Severity of URTI symptoms over the 84-day supplementation period. | baseline to day 84
  Severity of URTI symptoms over the 84-day supplementation period as determined by the average severity score of URTI symptoms. The average severity score of each symptom is scored on scale of 0- no symptom to 7-severe symptom. A higher score would indicate worse outcome.
The difference in proportion of participants with incidence of URTIs from day -14 to day -1. | day -14 to day -1
  The difference in proportion of participants with incidence of URTIs from day -14 to day -1 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
The difference in proportion of participants with incidence of URTIs from baseline to day 84. | baseline to day 84
  The difference in proportion of participants with incidence of URTIs from baseline to day 84 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
The difference in proportion of participants with incidence of URTIs from day -14 to day 84. | day -14 to 84
  The difference in proportion of participants with incidence of URTIs from day -14 to day 84 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
The difference in number of sick days from day -14 to day -1. | day -14 to day -1
  The difference in number of sick days from day -14 to day -1 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
The difference in number of sick days from baseline to day 84. | baseline to day 84
  The difference in number of sick days from baseline to day 84 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
The difference in number of sick days from day -14 to day 84. | day -14 to day 84
  The difference in number of sick days from day -14 to day 84 as assessed by the WURSS-24 questionnaire will be compared between Bio Gelee Royale Forte and Placebo.
Use of prescription and non-prescription cold/flu medications to treat URTI symptoms between day -14 to day -1. | day -14 to day -1
  Use of prescription and non-prescription cold/flu medications to treat URTI symptoms between day -14 to day -1 will be compared between Bio Gelee Royale Forte and Placebo.
Use of prescription and non-prescription cold/flu medications to treat URTI symptoms between baseline to day 84. | baseline to day 84
  Use of prescription and non-prescription cold/flu medications to treat URTI symptoms between baseline to day 84 will be compared between Bio Gelee Royale Forte and Placebo.
Use of prescription and non-prescription cold/flu medications to treat URTI symptoms between day -14 to day 84. | day -14 to day 84
  Use of prescription and non-prescription cold/flu medications to treat URTI symptoms between day -14 to day 84 will be compared between Bio Gelee Royale Forte and Placebo.

OTHER OUTCOMES:
Incidence of post-emergent adverse effects between day -14 to day 84. | day -14 to day 84
  Incidence of post-emergent adverse effects between day -14 to day 84.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, PhD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada